CLINICAL TRIAL: NCT02466308
Title: Long Duration Therapeutic Ultrasound for Tendon Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZetrOZ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TN-01
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2015-06

CONDITIONS: Tendinopathy; Tendinitis; Tendinosis
Keywords: sustained acoustic medicine; therapeutic ultrasound; SAM; LITUS
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SAM Ultrasound Diathermy Device (Experimental): SAM (sam Professional System) 3 MHz ultrasound diathermy device: 4 hours/day, at least 5 days per week, for 6 weeks
  Interventions: Device: SAM Ultrasound Diathermy Device

INTERVENTIONS:
Device: SAM Ultrasound Diathermy Device
  Other Names: sustained acoustic medicine; SAM

SUMMARY:
ZetrOZ's Ultrasonic Diathermy device (sam(R) Professional System) is intended for use as a portable and wearable medical device which, when applied to various areas of the body applies Low Intensity Therapeutic Ultrasound (LITUS) to deep tissues. This device is FDA-cleared for pain reduction, treatment of muscle spasm and joint contracture, and increasing local circulation. This study will look at the use of therapeutic ultrasound to relieve pain and enhance tendon extensibility for individuals with tendinopathy over a 6 week time period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18-65 years of age, inclusive
* Diagnosis of tendinitis in the elbow (lateral or medial epicondyle), Achilles tendon, or patellar tendon based on examination of medical history and confirmed by physical examination including either manual movements of the injured limb, e.g., a positive Mill's Test for elbow tendinitis, or local tenderness upon palpation of the tendon;
* Body mass index (BMI) less than or equal to 30.0
* Not taking NSAIDs or prescription pain medications for their tendinitis, and agree to document all pain medication use during the study period.

Exclusion Criteria:

* History or current diagnosis of tendon tear in treated tendon
* Known neuropathy
* Type I or Type II diabetes mellitus
* Had surgery in target treatment area within 6 months
* Refuse to agree to not increase current use or initiate new use of pain medication during the trial unless medically necessary to ensure patient safety
* Refuse to agree to not use any cream, gel, or topical solution during the administration of treatment other than the approved ultrasound gel provided
* Refuse to discontinue all other interventional treatment modalities (e.g., transcutaneous electrical nerve stimulation, other ultrasound therapy, etc.)
* Have had a local corticosteroid or platelet-rich plasma injection within the past 3 months
* Have participated in a clinical trial for an investigational drug and/or agent within 30 days prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Pain (Numeric Rating Scale; NRS) | Change from Baseline to Week 6

SECONDARY OUTCOMES:
Pain (NRS): 50% response rate | Week 6
Pain (NRS) during treatment session | Pre-treatment to Post-treatment (4 hours)
Grip Strength (dynamometer) | Change from Baseline to Week 6
Treatment Compliance (subject-reported use of device compared to protocol) | weekly through Week 6

CONTACTS AND LOCATIONS:
Locations (1):
- ZetrOZ, Inc., Trumbull, Connecticut, United States

REFERENCES:
- [Derived] Best TM, Moore B, Jarit P, Moorman CT, Lewis GK. Sustained acoustic medicine: wearable, long duration ultrasonic therapy for the treatment of tendinopathy. Phys Sportsmed. 2015 Nov;43(4):366-74. doi: 10.1080/00913847.2015.1095617. Epub 2015 Oct 15. PMID 26468991